CLINICAL TRIAL: NCT06610942
Title: Characterization of the Fungal Immunopeptidome Involved in the Immunopathological Mechanisms of Psoriasis
Acronym: PSOFUNGI
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240968; 2024-A01701-46 (Other: IDRCB ANSM)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis
Keywords: Fungi; immunopeptidome; psoriasis; IL17
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Adult patients with psoriasis who have failed local treatment
- "Healthy" controls (skin)
- "Healthy" controls (stools)

SUMMARY:
Psoriasis is a chronic immune-mediated skin disorder characterized by inflammatory cutaneous plaques and, occasionally, arthritis, affecting 60 million adults and children worldwide. Although a variety of treatments have been developed aimed to relieve the associated symptoms, there is yet no permanent cure for psoriasis. TH17 type immunity, via the production of IL-17A and other pro-inflammatory cytokines, are considered to play a central role in the pathogenesis of this disease. Moreover, experimental evidence obtained in animal models, points to human mycobiota as a trigger for the initiation and/or progression of psoriasis. Therefore, human studies are required to better characterize the major fungi implicated in the local and systemic inflammatory responses, as well as to determine the immunopeptidome that shapes the pathogenic T cell receptor repertoire.

We will explore the hypothesis that commensal fungi could participate in the chronic inflammatory immune response underlying the pathogenesis of human psoriasis via the recognition of cutaneous fungal antigens and/or via a gut-skin mycobiome cross-reactive mechanism

DETAILED DESCRIPTION:
The overall aim of the project is :

i) to characterize the nature of human local and systemic inflammatory responses against commensal skin and gut fungal species in psoriatic patients (PsoP) and ii) to determine the fungal immunopeptidome that contributes to the shaping of the T cell receptor (TCR) repertoire of skin-infiltrating T cells. The project is divided into four major scientific objectives:

1. To determine the mycobiome profiles in healthy donors (HD) and PsoP.
2. To characterize the contribution of mycobiota to the local cutaneous CD4+ T cell response.
3. To assess systemic the CD4+ T cell-fungal cross-reactivity.
4. To establish the immunopeptidome of the major CD4+ T cell-reactive fungus enabling the development of an innovative immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

Adults with psoriasis failing local treatment. Adults requiring reconstructive plastic surgery (resident skin immunology checks).

Adults living in the same household as a patient suffering from psoriasis (intestinal mycobiome checks).

Exclusion Criteria:

Minors Individuals under legal protection. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with psoriasis failing local treatment. Studying various biological samples from these patients (skin, blood, stools, and skin swabs) will allow the investigation of the local and systemic immune response and an attempt to understand the involvement of the skin and intestinal mycobiome.
  Healthy controls (skin): Adult patients undergoing reconstructive surgery where healthy skin is removed. Studying samples of healthy skin will enable the investigation of the skin immune response in subjects without skin disease or autoimmune disease.
  Healt controls (stools): Living in the same household as the patient with psoriasis. This population will allow the study of the intestinal mycobiome in controls with environments and diets similar to those of patients with psoriasis.
  Healthy controls (blood): Blood samples from donors obtained from the French Blood Establishment (EFS). These samples will allow the study of the systemic immune response to better understand the
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Determining the commensal fungi responsible for the immunopathological response in psoriasis. | 2 years
  Flow cytometry analysis of cytokine secretion profile in healthy and diseased subjects

SECONDARY OUTCOMES:
Identification of peptides responsible for the immunopathological response in psoriasis. | 2 years
  LC-MS/MS analysis of MHC I and II peptides

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Parasitologie-Mycologie Hôpital St Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No